CLINICAL TRIAL: NCT06283849
Title: Collaborative Solutions for Breaking up Sedentary Time in Black Older Adults With Type 2 Diabetes: The Interrupt Diabetes Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SON-2024-32671
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Explanatory sequential mixed methods study of N=30 Black adults aged 55 and older with T2D.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Black adults aged 55 and older with T2D
  Interventions: Behavioral: strategies to break up SB

INTERVENTIONS:
Behavioral: strategies to break up SB — Participants will be asked to implement strategies to break up their SB every hour for at least 8 hours a day for one week. Strategies will be developed through collaboration with participants during the first study interview and may include (but are not limited to): calf raises, brief (~5 min) self-paced walking), squats, sit to stand, etc. Participants will wear an activity monitor for assessment of SB and walking. This device (activPAL, PALTechnologies, Glasgow, Scotland) is not an investigational device; it is used for monitoring sedentary behavior.

SUMMARY:
The disparate burden of Type 2 Diabetes (T2D) faced by Black individuals makes attention to preventing or delaying the development of T2D and its associated cardiovascular (CV) complications, essential.

Similar to differences in cardiovascular disease (CVD) rates across racial and ethnic groups of older people, there are differences in engagement in physical activity (PA), a significant contributor to CVD. Black adults are less likely to engage in physical activity PA than their non-Hispanic White peers, with 26.7% of Black Minnesotans reporting that they did not engage any leisure-time PA in the past month, compared to 19.6% of non-Hispanic White Minnesotans. Notably, recent research has demonstrated that high amounts SB (i.e., sitting or lying with low levels of energy expenditure) also have significant detrimental effects on health, beyond those of physical inactivity. Experimental data from lab-based studies demonstrate that breaking up prolonged SB can rapidly improve markers of cardiometabolic risk (e.g., glucose and endothelial function) but the majority of these studies have focused on young, healthy, White adults. Given the significant inequities and health disparities faced by Black individuals and the lack of adequate representation of Black older adults in studies examining SB in individuals with T2D, understanding psychosocial and societal contributors to and consequences of SB experienced by this population is an essential first step toward developing relevant interventions targeting SB, and ultimately, CV health.

The disparate burden of T2D faced by Black individuals makes attention to preventing or delaying the development of T2D and its associated CV complications, essential.

Similar to differences in CVD rates across racial and ethnic groups of older people, there are differences in engagement in physical activity (PA), a significant contributor to CVD. Black adults are less likely to engage in PA than their non-Hispanic White peers, with 26.7% of Black Minnesotans reporting that they did not engage any leisure-time PA in the past month, compared to 19.6% of non-Hispanic White Minnesotans. Notably, recent research has demonstrated that high amounts SB (i.e., sitting or lying with low levels of energy expenditure) also have significant detrimental effects on health, beyond those of physical inactivity. Experimental data from lab-based studies demonstrate that breaking up prolonged SB can rapidly improve markers of cardiometabolic risk (e.g., glucose and endothelial function) but the majority of these studies have focused on young, healthy, White adults. Given the significant inequities and health disparities faced by Black individuals and the lack of adequate representation of Black older adults in studies examining SB in individuals with T2D, understanding psychosocial and societal contributors to and consequences of SB experienced by this population is an essential first step toward developing relevant interventions targeting SB, and ultimately, CV health.

The goal is to develop a deeper understanding of individuals' experiences of sedentary behavior (SB) and collaborate to design strategies to reduce SB. Using the Center for Chronic Disease Reduction and Equity Promotion Across Minnesota (C2DREAM) conceptual model, social-ecological framework, and COM-B model, the study will seek to understand the relationship between SB and individual, relationship, community, and societal factors. The study will also examine the context of SB and strategies that participants have used and could or would consider using to break up the time they spend sitting.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black or African American.
* Aged 55 years and older.
* Speak and read English.
* Self-reported diagnosis of T2D.

Exclusion Criteria:

* Evidence of cognitive impairment that could impact ability to consent and/or participation (Mini-Cog score <3).
* Physical impairment or disability that interferes with ability to engage in PA (e.g., severe osteoarthritis, lower extremity amputation [other than toe(s)/partial foot], regular use of a walker or wheelchair, etc.).
* Unstable medical/psychiatric condition that in the opinion of the PI could impact study participation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
sedentary time | 7 days
  measured via accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Mary O Whipple, PhD, RN, PHN, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States